CLINICAL TRIAL: NCT03826186
Title: Traditional Loss-of-resistance Technique vs Compuflo-aided Technology for Placement of a Thoracic Epidural Catheter: a Randomized Trial of the Effect on the Success Rate
Brief Title: CompuFlo Thoracic Epidural Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: YATISH SIDDAPURA RANGANATH (Other)
Responsible Party: Sponsor-Investigator, YATISH SIDDAPURA RANGANATH, Clinical Assistant Professor, University of Iowa
Organization: University of Iowa (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 201812716
Record Dates: First submitted 2019-01-22; First posted 2019-02-01 (Actual); Results first posted 2022-10-19 (Actual); Last update posted 2022-10-19 (Actual); Status verified 2022-08

CONDITIONS: Thoracic Epidural Anesthesia
Keywords: CompuFlo; dynamic pressure sensing

STUDY DESIGN:
Intervention Model Description: Thoracic epidurals are administered. After randomization, one group will receive thoracic epidurals in the traditional way (control group) and the other with CompuFlo assistance (study group).
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Traditional epidural group (Active Comparator): The traditional approach to placing thoracic epidurals by loss-of-resistance technique using a ground glass syringe will be used in this group.
  Interventions: Device: Traditional (loss-of-resistance technique) thoracic epidural placement
- CompuFlo epidural group (Experimental): This device (CompuFlo) will aid in correct placement of the epidural by electronically sensing pressure in real time and by providing a numerical value on a read out screen to determine a loss of resistance. There is also an audio signal that signals a loss of resistance.
  Interventions: Device: CompuFlo thoracic epidural placement

INTERVENTIONS:
Device: Traditional (loss-of-resistance technique) thoracic epidural placement — Thoracic epidurals will be administered using the traditional loss-of resistance technique.
  Arms: Traditional epidural group
Device: CompuFlo thoracic epidural placement — Pressure sensing technology to consistently and accurately identify the thoracic epidural space.
  Arms: CompuFlo epidural group

SUMMARY:
Traditionally, loss-of-resistance (LOR) to air or saline with a special ground-glass syringe is the technique used to identify epidural space, but failure rates up to 30% have been reported using this technique for thoracic epidural placement. This failure rate has sparked the search for newer techniques to improve the success rate for placement.The CompuFlo epidural system is a device that provides anesthesiologists and other healthcare providers the ability to quantitatively determine and document the pressure at the needle tip in real time. The device's proprietary dynamic pressure sensing technology (DPS) allows it to provide objective visual and audible in-tissue pressure feedback that allows anesthesiologists to identify the epidural space. The purpose this research study is to compare the success rate of the two different approaches (traditional method v/s CompuFlo assisted) to thoracic epidural placement.

DETAILED DESCRIPTION:
Traditional technique vs CompuFlo use: Using the traditional technique (loss-of-resistance technique), the epidural needle is advanced through the subcutaneous tissues with the needle stylet in place until the needle tip is positioned in the interspinous ligament-this is noted by the proceduralist by an increase in tissue resistance (attempted injection into ligamentous tissue is met with high resistance). The stylet or introducer is removed, and a ground-glass syringe filled with 2-3 mL of saline with an air bubble is attached to the hub of the epidural needle. If the tip of the needle is within the ligament, gentle attempts at injection are met with resistance, and injection of the saline is not possible. The needle is then slowly advanced, millimeter by millimeter, with either continuous or rapidly repeating attempts at injection. As the tip of the needle enters the posterior epidural space, a sudden loss of resistance is noted, and the saline injects easily. Once the needle tip is in the epidural space, the epidural catheter is threaded through the needle and the needle is removed, leaving the catheter sited in the epidural space.

The CompuFlo technique complements this basic technique. Similar to the traditional technique, the needle is advanced through the subcutaneous tissues with the stylet in place until the interspinous ligament is entered, as noted by an increase in tissue resistance. After removing the stylet, flexible tubing from the CompuFlo disposable tubing-syringe set is attached to the hub of the needle instead of the traditional ground-glass syringe. The fluid-filled syringe is placed in the CompuFlo device. The needle is then advanced continuously with the device electronically sensing pressure in real time, providing a numerical value (100 to 150 mm Hg) on the read-out screen. As the tip of the needle enters the posterior epidural space, a sudden loss of resistance (associated with a significant loss of pressure to less than 50 mm Hg or 50% of the starting pressure) is noted. The pressure drop needs to be sustained for at least 5 seconds. An audio signal also signals the acute change in pressure.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18 to 70
* BMI: 18 to 50 kg/m2
* Require pain control for major thoracic or abdominal surgeries
* Require pain control for rib fractures
* English is the subject's first language
* Must be able to signed informed consent

Exclusion Criteria:

* Age: Less than 18 and older than 70
* Must be free of significant valvular heart disease
* Pregnant women
* Prisoners
* Contraindication to thoracic epidural anesthesia
* Allergy or hypersensitivity to local anesthetics
* Unable to provide written informed consent

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2019-03-26 (Actual); Primary Completion 2022-01-01 (Actual); Study Completion 2022-06-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yatish S Ranganath, MD, Principal Investigator — University of Iowa
Locations (1):
- University of Iowa Hospitals and Clinics, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: Yes
All of the individual participant data (IPD) collected during the trial, after deidentification will be shared with researchers who provide a methodologically sound proposal, to achieve aims in the approved proposal. Individual participant data will be available for sharing immediately after publication and ending 5 years following article publication.
Supporting Information: Study Protocol, ICF
Time Frame: Individual participant data will be available for sharing immediately after publication and ending 5 years following article publication.
Access Criteria: Individual participant data will be accessible to researchers who provide a methodologically sound proposal, to achieve aims in the approved proposal.

REFERENCES:
- [Result] Block BM, Liu SS, Rowlingson AJ, Cowan AR, Cowan JA Jr, Wu CL. Efficacy of postoperative epidural analgesia: a meta-analysis. JAMA. 2003 Nov 12;290(18):2455-63. doi: 10.1001/jama.290.18.2455. PMID 14612482
- [Result] Carli F, Mayo N, Klubien K, Schricker T, Trudel J, Belliveau P. Epidural analgesia enhances functional exercise capacity and health-related quality of life after colonic surgery: results of a randomized trial. Anesthesiology. 2002 Sep;97(3):540-9. doi: 10.1097/00000542-200209000-00005. PMID 12218518
- [Result] Popping DM, Elia N, Marret E, Remy C, Tramer MR. Protective effects of epidural analgesia on pulmonary complications after abdominal and thoracic surgery: a meta-analysis. Arch Surg. 2008 Oct;143(10):990-9; discussion 1000. doi: 10.1001/archsurg.143.10.990. PMID 18936379
- [Result] Leurcharusmee P, Arnuntasupakul V, Chora De La Garza D, Vijitpavan A, Ah-Kye S, Saelao A, Tiyaprasertkul W, Finlayson RJ, Tran DQ. Reliability of Waveform Analysis as an Adjunct to Loss of Resistance for Thoracic Epidural Blocks. Reg Anesth Pain Med. 2015 Nov-Dec;40(6):694-7. doi: 10.1097/AAP.0000000000000313. PMID 26469364
- [Result] Parra MC, Washburn K, Brown JR, Beach ML, Yeager MP, Barr P, Bonham K, Lamb K, Loftus RW. Fluoroscopic Guidance Increases the Incidence of Thoracic Epidural Catheter Placement Within the Epidural Space: A Randomized Trial. Reg Anesth Pain Med. 2017 Jan/Feb;42(1):17-24. doi: 10.1097/AAP.0000000000000519. PMID 27922948
- [Result] Gong Y, Shi H, Wu J, Labu D, Sun J, Zhong H, Li L, Xin X, Wang L, Wu L, Ma D. Pressure waveform-guided epidural catheter placement in comparison to the loss-of-resistance conventional method. J Clin Anesth. 2014 Aug;26(5):395-401. doi: 10.1016/j.jclinane.2014.01.015. Epub 2014 Aug 27. PMID 25172504
- [Derived] Ranganath YS, Ramanujam V, Al-Hassan Q, Sibenaller Z, Seering MS, Singh TSS, Punia S, Parra MC, Wong CA, Sondekoppam RV. Loss-of-Resistance Versus Dynamic Pressure-Sensing Technology for Successful Placement of Thoracic Epidural Catheters: A Randomized Clinical Trial. Anesth Analg. 2024 Jul 1;139(1):201-210. doi: 10.1213/ANE.0000000000006792. Epub 2024 Jun 17. PMID 38190338

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Traditional Epidural Group | CompuFlo Epidural Group
Started | 60 | 60
Completed | 57 | 60
Not Completed | 3 | 0
Not completed — Protocol Violation | 2 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Traditional Epidural Group | CompuFlo Epidural Group | Total
Number analyzed (Participants) | 57 | 60 | 117
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.9 (11.34) | 57.9 (11.38) | 57.9 (11.36)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 35 | 65
  Male | 27 | 25 | 52
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 57 | 60 | 117

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Successful Thoracic Epidural Catheter Placement
Description: Successful placement of thoracic epidural analgesia will be determined by the loss of cold sensation on the chest or abdomen depending on the site of epidural placement using a dermatome bilaterally. Subjects will be tested at 10 minute intervals.
Time Frame: Maximum 20 minutes post administration of epidural test dose
Measure: Count of Participants; unit: Participants
Arm/Group | Traditional Epidural Group | CompuFlo Epidural Group
Number analyzed (Participants) | 57 | 60
Participants | 52 | 58

2. Secondary Outcome: Amount of Time Required to Complete the Procedure
Description: Tuohy needle skin puncture to removal of tuohy (for the last time) from the patient
Time Frame: During procedure, assessed up to 15 minutes
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Traditional Epidural Group | CompuFlo Epidural Group
Number analyzed (Participants) | 57 | 60
minutes | 8.02 (7.4) | 7.4 (6.6)

3. Secondary Outcome: Number of Participants Who Reported Loss of Cold Sensation at Various Time Points
Description: Record the time it takes for loss of cold sensation on the chest or abdomen depending on the site of epidural placement using a dermatome bilaterally. Subjects will be tested at 10 minute intervals.
Time Frame: Up to 20 minutes post administration of epidural test dose
Measure: Number; unit: participants
Arm/Group | Traditional Epidural Group | CompuFlo Epidural Group
Number analyzed (Participants) | 57 | 60
participants
  Loss of cold sensation-10 minutes | 28 | 18
  Loss of cold sensation-20 minutes | 24 | 40
  No change in cold sensation | 5 | 2

4. Secondary Outcome: Mean Arterial Pressure at Baseline and 20 Minutes Post Procedure
Description: Blood pressure was measured at baseline (patient check-in) and then every 5 minutes after administration of test dose in both groups. To observe the trend in blood pressure changes, the mean arterial pressure was used. Results are reported as mean arterial pressure (MAP) since MAP is the average arterial pressure throughout one cardiac cycle, systole and diastole. The MAP was calculated based on the available MAP formula (MAP=diastolic blood pressure (DBP) + 1/3 [systolic blood pressure (SBP) - DBP]).
Time Frame: Up to 20 minutes post administration of epidural test dose
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Traditional Epidural Group | CompuFlo Epidural Group
Number analyzed (Participants) | 57 | 60
mmHg
  Pre-procedure (mmHg) | 102 (14) | 102 (11)
  20-minutes after initial test dose | 85 (16) | 83 (14)

5. Secondary Outcome: Number of Participants With Significant Change in Systolic Blood Pressure
Description: A fall in systolic blood pressure by 20% or more from the baseline up to 20 minutes after the initial test dose was considered a significant change.
Time Frame: Up to 20 minutes post administration of epidural test dose
Measure: Count of Participants; unit: Participants
Arm/Group | Traditional Epidural Group | CompuFlo Epidural Group
Number analyzed (Participants) | 57 | 60
Participants | 41 | 38

6. Secondary Outcome: Number of Participants Whose Provider Answered "Yes" or "No" to Ease of Catheter Placement
Description: The provider was asked to evaluate the ease of catheter threading through the needle after the loss of resistance. This is a "yes" or "no" evaluation asked and answered at the end of the procedure. The question asked was "Was the catheter placement (threading) smooth after loss of resistance?"
Time Frame: During procedure, assessed up to 15 minutes
Measure: Number; unit: participants
Arm/Group | Traditional Epidural Group | CompuFlo Epidural Group
Number analyzed (Participants) | 57 | 60
participants
  Yes | 57 | 60
  No | 0 | 0

7. Secondary Outcome: Number of Participants With a Positive Meniscus Test
Description: The test involves 3 steps after removal of the filter: (i) the open end of the epidural catheter is lifted and the liquid meniscus present in the catheter is observed to drop rapidly; (ii) the open end of the epidural catheter is lowered and the liquid meniscus is again observed to fill the catheter with clear liquid and no blood; (iii) the presence of air in the catheter during backflow confirms the correct position in the epidural space relative to a position in the subarachnoid space. If the above changes are observed - that would help in secondary confirmation of the epidural space and we would call that a positive test. If the above changes are not observed, it was called as a negative test.
Time Frame: During procedure, assessed up to 15 minutes
Measure: Count of Participants; unit: Participants
Arm/Group | Traditional Epidural Group | CompuFlo Epidural Group
Number analyzed (Participants) | 57 | 60
Participants
  Positive | 57 | 57
  Negative | 0 | 3

8. Secondary Outcome: Number of Participants With Unintentional Dural Puncture
Description: The number of unintentional dural punctures during the traditional loss-of-resistance methods will be compared to the unintentional dural punctures while using the CompuFlo assisted technology.
Time Frame: During procedure, assessed up to 15 minutes
Measure: Count of Participants; unit: Participants
Arm/Group | Traditional Epidural Group | CompuFlo Epidural Group
Number analyzed (Participants) | 57 | 60
Participants | 2 | 2

ADVERSE EVENTS:
Time Frame: The data was collected from the time of consent until 48 hours post procedure.
Arm/Group | Traditional Epidural Group | CompuFlo Epidural Group
All-Cause Mortality (participants affected / at risk) | 0/57 | 0/60
Serious Adverse Events (participants affected / at risk) | 0/57 | 0/60
Other Adverse Events (participants affected / at risk) | 0/57 | 0/60

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol (2019-11-15): https://cdn.clinicaltrials.gov/large-docs/86/NCT03826186/Prot_003.pdf
  • Statistical Analysis Plan (2019-11-15): https://cdn.clinicaltrials.gov/large-docs/86/NCT03826186/SAP_004.pdf
  • Informed Consent Form (2019-11-15): https://cdn.clinicaltrials.gov/large-docs/86/NCT03826186/ICF_005.pdf